CLINICAL TRIAL: NCT01116180
Title: Influence of Blockade of the Renin-angiotensin System for Preservation of Cognitive Function, Hormonal Counter-regulatory Response, Symptomatology and Cardiac Repolarisation During Hypoglycaemia in Patients With Type 1 Diabetes
Brief Title: Cognitive Function and Electrocardiogram (ECG) During Hypoglycemia and Blockade of the Renin-angiotensin System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louise Faerch (Other)
Responsible Party: Sponsor-Investigator, Louise Faerch, MD, ph.d.student, Hillerod Hospital, Denmark
Organization: Hillerod Hospital, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HypoRas
Record Dates: First submitted 2010-01-25; First posted 2010-05-04 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Type 1 diabetes; Hypoglycaemia; genetic susceptibility; Renin angiotensin system activity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Genetic Predisposition to Disease | interventions — Angiotensin Receptor Antagonists; candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candesartan (Active Comparator)
  Interventions: Drug: Angiotensin II receptor antagonists (Candesartan)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Angiotensin II receptor antagonists (Candesartan) — Seven days of treatment with Candesartan 32 mg, capsules.
  Other Names: Blopress; Atacand; Amias; Ratacand
  Arms: Candesartan
Drug: Placebo — Placebo Capsule matching the active comparator. Given for 7 days once daily.
  Arms: Placebo

SUMMARY:
Hypothesis: Treating patients with type 1 diabetes with a certain antihypertensive drug preserve cerebral function during hypoglycaemia.

Background: Studies have found that certain genetic variations leaves a subject with type 1 diabetes more prone to hypoglycaemia. It it thought to be a decline in cognition during hypoglycaemia that leaves them at risk of severe hypoglycaemia. The idea is tha when you suppress the genetic phenotype with a well known antihypertensive drug an improvement in cognition will occur and this will remove the patients tendency to severe hypoglycaemia.

Methods: The investigators want to explore whether the cerebral function is improved during hypoglycaemia in subjects with type 1 diabetes and the above mentioned genetic variation when treated with the antihypertensive drug Candesartan.

DETAILED DESCRIPTION:
We will include 25 type 1 diabetic patients from our outpatient clinic. They are already genotyped from another trial.

Each patient goes through two cycles with hyperinsulinemic glucose clamp induced hypoglycemia. The study is double blinded, randomised and placebocontrolled so the patients receive both Candesartan and placebo but in different cycles.

In each cycle patients will receive either Candesartan or placebo for 7 days. After 8 days patients undergo a hypoglycaemic clamp during which primary and secondary endpoints will be measured.

In the hyperinsulinemic hypoglycaemic clamp the patients will undergo an adjustment period towards euglycaemia. A period of approximately 1 hour of euglycemia, an hour of hypoglycemia and a period of recovery towards euglycemia. In each of these glycemic states primary and secondary outcomes will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Danish spoken and written
* RAS activity score>7 - diabetes duration > 5 years
* not pregnant and safe anticonception
* Signed informed consent.

Exclusion Criteria:

* Treatment with an ACE blocker
* An ARB og a renin blocker
* Treatment with other antihypertensive drugs
* Severe diabetic late complications
* Renal impairment
* Pregnancy and breastfeeding
* Previous reactions to study medication
* Heart insufficiency (NYHA 3-4)\
* Known ischaemic heart disease
* Epilepsy
* Alcohol and drug abuse
* Suspicion of non-compliance,
* Plasma potassium < 3.5 mmol/l or >5.0 mmol/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Cognitive function and brain cortical activity assessed by EEG | 2 month

SECONDARY OUTCOMES:
Symptoms of hypoglycaemia assessed by Edinburgh Hypoglycaemia Symptom Score questionnaire | 2 month
Hormonal counter-regulatory response and substrates | 2 month
Blood pressure and pulse | 2 month
Cardiac conduction evaluated by a three channel digital Holter Monitor. | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Pedersen-Bjergaard, MD, MDSc., Study Director — Hillerød Hospital, Department of Cardiology and Endocrinology, Dyrehavevej 29, 3400 Hillerød; Louise Færch, MD, Principal Investigator — Hillerød Hospital, Department of Cardiology and Endocrinology, Dyrehavevej 29, 3400 Hillerød; Birger Thorsteinsson, Prof DMSc MD, Study Director — Hillerød Hospital, Department of Cardiology and Endocrinology, Dyrehavevej 29, 3400 Hillerød. University of Copenhagen
Locations (1):
- Department of Cardiology and Endocrinology, Hillerød Hospital, Hillerød, Denmark